CLINICAL TRIAL: NCT05700955
Title: A Phase I Trial of Neoadjuvant Chemoimmunotherapy in Recurrent Glioblastoma
Brief Title: Neoadjuvant Chemoimmunotherapy in Recurrent Glioblastoma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Louisville (Other)
Responsible Party: Principal Investigator, Donald Miller, Donald M. Miller, M.D., Ph.D., University of Louisville
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22.0676
Record Dates: First submitted 2022-09-28; First posted 2023-01-26 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — pembrolizumab; Temozolomide

STUDY DESIGN:
Intervention Model Description: The experience with neoadjuvant immunotherapy has raised the possibility of utilizing surgical resection/immunotherapy as a combination treatment for patients with recurrent glioblastoma. There are several reasons that suggest that surgical resection will likely enhance the activity of immunotherapy in glioblastoma.This includes 1) direct impact on tumor cells; 2) impact on immune cells; and 3) impact on immune infiltration. The combination of the evidence that neoadjuvant Pembrolizumab has a positive effect on GBM survival, the evidence in lung cancer that chemotherapy and checkpoint inhibitor therapies are synergistic and the clinical utility of surgery in patients with recurrent glioblastoma has suggested that the neoadjuvant administration of Pembrolizumab and temozolomide prior to and following maximal surgical resection represents a very attractive experimental combination for the treatment of recurrent glioblastoma.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- temozolomide (Experimental): Participants will take Temozolomide pills at home at a dose determined by body weight. They will take the pills for five days every 3 weeks. It will be dispensed by the pharmacy and must be stored in a closed container at room temperature, away from heat, moisture, and direct light and kept from freezing. It will be kept out of the reach of children. Outdated medicine or medicine no longer needed will be returned to the Brown Cancer Center pharmacy for disposal.
  Interventions: Drug: Pembrolizumab and Temozolomide
- Pembrolizumab (Experimental): Pembrolizumab will be administered at a dose of 200 mg as an IV infusion through a freely flowing IV. The diluted solution will be administered intravenously over 30 minutes through an intravenous line containing a sterile, non-pyrogenic, low-protein binding 0.2 micron to 5 micron in-line or add-on filter. Other drugs will not be co-administered through the same infusion line. Pembrolizumab doses will be repeated every three weeks.
  Interventions: Drug: Pembrolizumab and Temozolomide

INTERVENTIONS:
Drug: Pembrolizumab and Temozolomide — Characterize the safety and immunologic/genomic/metabolomic effects of neoadjuvant Pembrolizumab and Temozolomide in recurrent glioblastoma.
  Other Names: Pembro and Temodar

SUMMARY:
The primary purpose of this study is to test the safety of Pembrolizumab and Temozolomide in treating recurrent glioblastoma and to characterize the effect of this treatment on the participants tumor and immune system..

DETAILED DESCRIPTION:
Participants will undergo screening tests to determine if they are eligible to participate. This will involve a complete history and physical examination, vital signs, blood tests including complete blood count (CBC), and serum chemistry (CMP).

Participants will receive one cycle of Temozolomide and Pembrolizumab prior to removing recurrent tumor, followed by three weekly cycles of treatment until progression.

ELIGIBILITY:
Inclusion Criteria:

-Inclusion Criteria Patients are eligible to be included in the only if they meet all of the following criteria

1. Histopathologically proven diagnosis of glioblastoma prior to registration, by pathology report;
2. The tumor must be confined to the supratentorial compartment
3. The tumor tissue block from the primary diagnosis must be available to be sent for pathology review, after registration.
4. History/physical examination within 7 days prior to registration
5. Karnofsky performance status ≥ 60 within 7 days prior to registration.
6. Adequate Organ Function Laboratory Values

   * Absolute neutrophil count (ANC) ≥1,500/mcL
   * Platelets ≥100,000/mcL
   * Hemoglobin ≥9.0 g/gL or ≥5.6 mmol/L, without recent transfusion
   * Creatine ≤1.7 x upper limit of normal (ULN) or Measure or Calculated creatinine clearance ≥ 60.0mL/min for subject with creatinine levels > 1.5 X institutional ULN (GFR can also be used in place of creatinine or CrCl)
   * Total bilirubin ≤ 1.5 x ULN or Direct bilirubin ≤ ULN for subjects with total bilirubin levels > 1.5 x ULN
   * AST (SGOT) and ALT (SGPT) ≤ 2.5 x ULN or ≤ 5 x ULN for subjects with liver metastases
7. The patient must have completed chemoradiation with Radiotherapy and Temozolomide of the primary tumor according to standard of care.
8. Patients must have received no more than 3 prior therapies for Recurrent High Grade Glioma.
9. Subjects must have the ability to understand and willingness to sign a written informed consent document.
10. Female subjects of childbearing potential should have a negative urine or serum pregnancy test within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
11. Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication.
12. Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy.

Exclusion Criteria:

-Exclusion Criteria Patients will be excluded from the study if they meet any of the following criteria

1. Previous use of an immunotherapy such as a vaccine therapy, dendritic cell vaccine or intracavitary or convectional enhanced delivery of therapy.
2. Prior invasive malignancy (except non-melanomatous skin cancer) within the previous three years
3. Severe, active co-morbidity defined as follows:

   * Transmural myocardial infarction or unstable angina within the last 6 months prior to registration
   * History of stroke, cerebral vascular accident (CVA) or transient ischemic attack within 6 months prior to registration
   * Significant vascular disease (e.g., aortic aneurysm, history of aortic dissection) or clinically significant peripheral vascular disease
   * Known history of Tuberculosis or acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration
   * Chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy at the time of registration
   * Patients with active autoimmune disease or history of autoimmune disease that might recur, will be considered on an individual basis
   * Any other major medical illnesses or psychiatric impairments that in the investigator's opinion will prevent administration or completion of protocol therapy.
   * Is pregnant or breastfeeding
   * Has received prior therapy with an anti-Programmed Death 1 (PD-1), anti- Programmed Death-ligand 1 (PD-L1), or anti- Programmed Death-ligand 1 (PD-L2) agent.
4. Patient must have < 1.5 cm midline shift pre-operative
5. History of severe hypersensitivity reaction to any monoclonal antibody including pembrolizumab.
6. Patients who cannot safely undergo MRI due to non-MRI compatible pacemaker, or other reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Treatment toxicity | Change in frequency of adverse events prior to gross total resection or recurrent glioblastoma
  Quantification of the frequency of adverse events in patients treated with neoadjuvant Pembrolizumab and Temozolomide with gross total resection of recurrent glioblastoma.

SECONDARY OUTCOMES:
Overall Survival | Every 8 weeks for 24 months
  Progression and response to treatment will be determined using the Response Assessment in Neuro-Oncology (RANO) criteria.
Neurologic function and quality of life | Every 8 weeks for 24 months
  Using the Neurologic Assessment in Neuro-oncology (NANO) scale on each visit. In addition, the Eastern Cooperative Oncology Group (ECOG) performance status will be monitored.
Treatment Toxicity | Change in frequency of adverse events after gross total resection or recurrent glioblastoma
  Quantification of the frequency of adverse events in patients treated with neoadjuvant Pembrolizumab and Temozolomide after gross total resection of recurrent glioblastoma.

CONTACTS AND LOCATIONS:
Overall Officials: Donald Miller, MD, Principal Investigator — University of Louisville/James Graham Brown Cancer Ctr.
Locations (1):
- James Graham Brown Cancer Ctr., Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No